CLINICAL TRIAL: NCT01170273
Title: Vitamin D in Vulnerable Adults
Brief Title: Vitamin D in Vulnerable Adults (VIVA-VA)
Acronym: VIVA-VA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: F7574-R
Record Dates: First submitted 2010-07-22; First posted 2010-07-27 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-10

CONDITIONS: Frail Elderly; Vitamin d Deficiency
Keywords: aged; vitamin d deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Arm (Placebo Comparator): placebo capsule
  Interventions: Dietary Supplement: placebo
- Cholecalciferol 4000 IU (Experimental): cholecalciferol 4000 IU daily
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D — cholecalciferol
  Arms: Cholecalciferol 4000 IU
Dietary Supplement: placebo — placebo tablet
  Arms: Placebo Arm

SUMMARY:
Vitamin D insufficiency is a problem of growing concern, given its prevalence in older persons and the association of low vitamin D with multiple major health problems, including mobility and balance deterioration and falls, cardiovascular disease, diabetes, and certain cancers. Sedentary persons are particularly vulnerable for these health problems and generally not adherent to prescribed physical activity. This study will investigate if treatment with vitamin D will benefit physical performance in male veterans age 65 to 95.

ELIGIBILITY:
Inclusion Criteria:

* male veterans
* 65 to 95 years of age
* independent
* sedentary
* vitamin D insufficiency

Exclusion Criteria:

* hypercalcemia
* renal failure
* living in a nursing home

Ages: 65 Years to 95 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-08; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvina Levis-Dusseau, MD, Principal Investigator — VA Medical Center, Miami
Locations (1):
- VA Medical Center, Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Arm: placebo capsule
  placebo: placebo tablet
  participants received one daily tablet containing placebo for 9 months
- Cholecalciferol 4000 IU: cholecalciferol 4000 IU daily
  vitamin D: cholecalciferol
  participants received one daily tablet containing cholecalciferol 4000 IU for 9 months
Period: Overall Study
Arm/Group | Placebo Arm | Cholecalciferol 4000 IU
Started | 64 | 66
Completed | 56 | 57
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 6 | 8
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Cholecalciferol 4000 IU | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (7.3) | 71.8 (6.3) | 72.4 (6.8)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 64 | 66 | 130

OUTCOME MEASURES:

1. Primary Outcome: Change in Short Physical Performance Battery Test Score
Description: The short physical performance battery (SPPB) examines 3 areas of lower extremity function: static balance test, gait speed test and getting in and out of a chair test. The total SPPB score is the sum of the scores of the 3 components and can range from 0 to 12, with 0 reflecting severe limitations and 12 minimal or no limitations. The ranges for each subscale are: balance (0-4), gait speed (0-4), sit-to-stand (0-4). In all the subscales, 0 reflects worse outcome and 4 best outcome.
Time Frame: baseline and 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Cholecalciferol 4000 IU
Number analyzed (Participants) | 56 | 57
units on a scale | 7.3 (1.69) | 7.0 (1.62)

ADVERSE EVENTS:
Arm/Group | Placebo Arm | Cholecalciferol 4000 IU
Serious Adverse Events (participants affected / at risk) | 5/64 | 2/66
Other Adverse Events (participants affected / at risk) | 12/64 | 11/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=64) | Cholecalciferol 4000 IU (N=66)
cancer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
pulmonary edema (Cardiac disorders) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
prostate cancer (Renal and urinary disorders) | 1 (1) | 0 (0)
lung cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Arm (N=64) | Cholecalciferol 4000 IU (N=66)
hypercalcemia (Endocrine disorders) | 1 | 3
fall (Injury, poisoning and procedural complications) | 11 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes